CLINICAL TRIAL: NCT02038634
Title: Ultrasound-guided Injection for DeQuervain's
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: not enough patient data
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Steven Grindel, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO20646
Record Dates: First submitted 2013-09-25; First posted 2014-01-16 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: DeQuervain's Tenosynovitis
Keywords: wrist; tendonitis; dequervain's; tenosynovitis
MeSH Terms: conditions — Tendinopathy; Tenosynovitis | interventions — Betamethasone; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unguided injections (Active Comparator): Corticosteroid injection (betamethasone) without ultrasound guidance.
  Interventions: Drug: Betamethasone
- Ultrasound-guided injections (Active Comparator): Corticosteroid injections (betamethasone) under ultrasound guidance.
  Interventions: Drug: Betamethasone; Device: Ultrasound

INTERVENTIONS:
Drug: Betamethasone
  Other Names: celestone
Device: Ultrasound — Ultrasound guided injection using GE Healthcare LOGIQ e Ultrasound
  Arms: Ultrasound-guided injections

SUMMARY:
The investigators aim to perform a prospective study to evaluate the effectiveness of blind corticosteroid injections to US-guided injections for the treatment of de Quervain's disease. The results of the study will be used to validate current injection protocols or support the incorporation of ultrasonography to treat the disease.

DETAILED DESCRIPTION:
De Quervain's disease is the stenosing tenosynovitis and tendinitis of the abductor pollicis longus (APL) and extensor pollicis brevis (EPB) tendons in the first dorsal compartment of the wrist. While the prevalence of de Quervain's is not yet well-established, previous studies have shown that women can be affected by the disease up to six times more frequently than men. Conservative treatments include splinting and corticosteroid injections, but surgery is an option when such therapy fails. There has been a previous study that compared the improvement rates of patients treated with splinting alone, injection and splinting, and injection alone, and found the rate of improvement to be 19%, 57%, 67%, respectively. This confirmed the good results reported in previous studies and recommends corticosteroid injection to clinicians as a reliable treatment for de Quervain's disease.

A seminal study performed correlated the accuracy of corticosteroid injection with pain relief by including X-ray dye in the injection. The results of the study suggested a strong correlation between accurate injection of the first dorsal compartment and pain relief. Since then, the use of ultrasonography (US) to guide steroid injection has been suggested as a possible clinical practice, but little research has been done on the technique. A 2009 study reported a 93.75% rate of significant pain relief after the use of US-guided injections, but there was no control group with which to compare results. The current standard practice for steroid injection in de Quervain's patients is a blind injection without imaging guidance. To the investigators knowledge, no study has compared the accuracy and clinical outcomes of blind injections to US-guided injections. The investigators hypothesize that the US-guided injections will be and will result in greater pain relief for patients than blind injections.

This is intended to be a prospective study. Patients will contact Dr.'s Grindel and Daley for a standard clinical evaluation, which includes palpation of the first extensor compartment and application of the Finkelstein test. Those diagnosed with de Quervain's disease and who fit all inclusion criteria will receive a detailed verbal description of the study from one of the doctors, who will then attain written, informed consent from willing participants. Dr.'s Grindel or Daley will then administer either a blind or US-guided injection. The patient will return for follow-up appointments at 6-8 weeks and 12-16 weeks and will undergo another physical exam to determine pain relief. A phone call follow-up will also be placed one year after the injection in order to determine long-term effectiveness. Once 20 study subjects in each group (40 total) have been enrolled and completed treatment, the data will undergo statistical analysis.

This study poses minimal or no physical risk to study subjects, as the US-guided injection should show better pain relief for patients than the current standard treatment (blind injection).

In summary, the investigators aim to perform a prospective study to evaluate the effectiveness of blind corticosteroid injections to US-guided injections for the treatment of de Quervain's disease. The results of the study will be used to validate current injection protocols or support the incorporation of ultrasonography to treat the disease.

ELIGIBILITY:
Inclusion Criteria:

* Pain with palpation at 1st dorsal compartment at wrist and positive Finkelstein's Test

Exclusion Criteria:

* Patients with evidence of osteoarthritis or degeneration of the wrist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grindel, MD, Principal Investigator — MCW/Froedtert Hospital
Locations (1):
- Froedtert Hospital, Wauwatosa, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
We have no plan to share the data we have collected with any other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based by the PI between August 2013 and April 2021. The first participant was enrolled on August 5, 2014 and the last participant was enrolled on December 9, 2018
Pre-assignment Details: 16 met inclusion criteria and were randomized to treatment.
Groups:
- Unguided Injections: Corticosteroid injection (betamethasone) without ultrasound guidance.
  Betamethasone
- Ultrasound-guided Injections: Corticosteroid injections (betamethasone) under ultrasound guidance.
  Betamethasone
  Ultrasound: Ultrasound guided injection using GE Healthcare LOGIQ e Ultrasound
Period: Overall Study
Arm/Group | Unguided Injections | Ultrasound-guided Injections
Started | 3 | 13
Completed | 3 | 12
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unguided Injections | Ultrasound-guided Injections | Total
Number analyzed (Participants) | 3 | 13 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 11 | 13
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 13 | 15
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: DASH - "Disabilities of the Arm, Shoulder, and Hand" Score At Baseline, and Change From Baseline at 6-8 Weeks, 12-16 Weeks, and at 1 Year
Description: Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire. Questions 1-30, the scale is a 1-5 scale (1=no difficulty; 2=mild difficulty; 3=moderate difficulty; 4=severe difficulty; 5=unable) DASH Disability/Symptom Score = [(sum of n responses)/n) -1] x 25. A lower score is a better outcome. The Dash is based on a scale of 0-100. Our scores were averaged and the Mean scores are what we reported. Total scores are listed below.
  US Guided Group - Dash #1 (Min=25, Mean=58, Max=90) n=12; Dash #2 (Min=3, Mean=38, Max=91) n=12; Dash #3 (Min=6, Mean=42, Max=71) n=10; 1 Year Dash (Min=0, Mean =29, Max=91) n=12.
  Non-US Guided Group - Dash #1 (Min=23, Mean=39, Max=61) n=3; Dash #2 (Min=0, Mean=11, Max=22) n=3; Dash #3 (Min=7, Mean=30, Max=49) n=3; 1 Year Dash (Min=0, Mean=9, Max=25) n=3.
Time Frame: Prior to injection (Dash #1), 6-8 weeks (Dash #2), 12-16 weeks (Dash #3), and 1 year (Dash #4) post-injection
Population: We enrolled 3 subjects into the Unguided Injection Arm and 13 subjects into the Ultrasound-Guided Injection Arm, however no further data was analyzed due to early termination of study.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Unguided Injections | Ultrasound-guided Injections
Number analyzed (Participants) | 3 | 13
score on a scale
  Dash #1 Pre-Injection: number analyzed (Participants) | 3 | 12
  Dash #1 Pre-Injection | 39 [23 to 61] | 58 [25 to 90]
  Dash #2 6-8 Weeks: number analyzed (Participants) | 3 | 12
  Dash #2 6-8 Weeks | 11 [0 to 22] | 38 [3 to 91]
  Dash #3 12-16 Weeks: number analyzed (Participants) | 3 | 10
  Dash #3 12-16 Weeks | 30 [7 to 49] | 42 [6 to 71]
  Dash #4 - 1 Year: number analyzed (Participants) | 3 | 12
  Dash #4 - 1 Year | 9 [0 to 25] | 29 [0 to 91]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 1 year.
Arm/Group | Unguided Injections | Ultrasound-guided Injections
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/13
Other Adverse Events (participants affected / at risk) | 0/3 | 0/13

LIMITATIONS AND CAVEATS:
Early termination due to lack of subject participation; statistical analysis not done due to small numbers. Outcome Measure # 2 was originally posted but was deleted as it was not included as part of the study design. No data was collected for that proposed outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT02038634/Prot_SAP_000.pdf